CLINICAL TRIAL: NCT05279560
Title: The Efficacy and Safety of Intra-ovarian PRP Injection Within a Prospective, Single-blinded, Placebo-controlled, Randomized, Clinical Superiority Trial in Subjects With Low Ovarian Reserve/Expected Poor Ovarian Response
Brief Title: Ovarian PRP (Platelet Rich Plasma) Injection for Follicular Activation
Acronym: OPIF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Luebeck (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. M.Sc. Georg Griesinger, Head of Department of Gynecological Endocrinology and Reproductive Medicine, University of Luebeck
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Aktenzeichen 21-348
Record Dates: First submitted 2022-01-16; First posted 2022-03-15 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Premature Ovarian Insufficiency; Infertility, Female; Sterility, Female; PRP
Keywords: poor ovarian response; low ovarian response; ICSI; IVF; ART; Platelet rich plasma; PRP
MeSH Terms: conditions — Primary Ovarian Insufficiency; Infertility, Female | interventions — Saline Solution; Injections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autologous intra-ovarian PRP injection (Experimental): Study group, treated with autologous intra-ovarian PRP injection and undergoing a subsequent fresh ET-IVF/ICSI cycle in the third cycle after intervention
  Interventions: Biological: autologous PRP (platelet rich plasma)
- intra-ovarian saline solution (NaCL) injection (Placebo Comparator): Control group, treated with intra-ovarian NaCl injection and undergoing a subsequent fresh ET-IVF/ICSI cycle in the third cycle after intervention
  Interventions: Other: Saline solution (NaCL) Injection

INTERVENTIONS:
Biological: autologous PRP (platelet rich plasma) — The required volume of PRP will be extracted from 60 ml of the patient's peripheral blood. Injecting PRP into the ovaries will be performed likewise to the standard operating procedure of oocyte retrieval. After centrifugation of the whole blood, 5ml PRP will be injected in each ovary intra-medullar and subcortical using a 17-gauge single lumen needle under sedation und under transvaginal ultrasound monitoring.
  Arms: Autologous intra-ovarian PRP injection
Other: Saline solution (NaCL) Injection — Injecting NaCL into the ovaries will be performed likewise to the standard operating procedure of oocyte retrieval. NaCL will be injected in each ovary intra-medullar and subcortical using a 17-gauge single lumen needle under sedation und under transvaginal ultrasound monitoring.
  Arms: intra-ovarian saline solution (NaCL) injection

SUMMARY:
The primary objective is to investigate the efficacy, defined as an increase in oocyte numbers upon ovarian stimulation, and safety of a single intra-ovarian PRP injection vs. saline solution (NaCl) injection (Placebo) transvaginally or laparoscopically for follicular activation in patients with child wish and with low ovarian reserve/expected poor ovarian response planning to undergo IVF or ICSI using own eggs. Pain score as numerical rating score and validated quality of life questionnaire will be requested after the procedure. Longterm follow-up of all participants will be performed 1, 2 and 5 years after end of study.

DETAILED DESCRIPTION:
Age-related infertility and premature loss of ovarian reserve has become a major challenge for ART professionals as the the average age at first child wish has dramatically increased over time. Under physiological circumstances, most follicles in the human ovary remain dormant throughout the female life span and eventually become atretic, however, histological samples reveal that the follicular pool in the ovary is completely exhausted only as late as the early 70ies and that the ovary holds oogonial stem cells, which may have the ability to differentiate into functional follicles. The pressing problem for reproductive medicine is therefore the question how to reactivate some of the putative ovarian 'reproductive reserve' in those women with premature follicular depletion or those who wish to become pregnant at advanced age.

Platelet rich plasma (PRP) is a blood-derived product, characterized by high concentrations of growth factors and chemokines. PRP is produced by centrifuging a small quantity of the patient's own blood and extracting the active, platelet-rich fraction. The platelet-rich fraction is applied to the human body typically by injection. PRP is used for therapeutic purposes in different medical areas ranging from orthopedics to plastic surgery, for its putative ability to stimulate and facilitate cell proliferation and thereby tissue differentiation and regeneration.

In the context of reproductive medicine, PRP has been proposed to increase pregnancy rates after uterine flushing in women with recurrent implantation failure or thin endometrium. Intra-ovarian injection of PRP has been proposed to activate dormant ovarian follicles pre IVF-treatment in cases of idiopathic low ovarian reserve, premature ovarian insufficiency or ovarian depletion because of advanced maternal age. To date, there is no randomized placebo-controlled trial available that has evaluated intra-ovarian PRP injection in terms of efficacy and safety for premature ovarian failure, and, more specifically, also not in patients with depleted ovarian reserve/poor ovarian response (POR) who constitute a significant proportion of patients undergoing assisted reproduction.

ELIGIBILITY:
Inclusion Criteria:

* Serum AMH < 0.5 ng/ml (at screening visit and in the absence of OC or sex-steroid intake)
* Antral follicular count (AFC) in both ovaries ≤ 5 (at screening visit and in the absence of OC or sex-steroid intake)
* Spontaneous cycle, menstrual cycle length 21-35 days
* Body mass index (BMI) ≥18 kg/m2 and ≤38 kg/m2
* Both ovaries must be visible by transvaginal ultrasound examination
* Both ovaries must be judged accessible by transvaginal puncture
* Indication for IVF or ICSI treatment
* Willingness to participate and provide written consent prior to initiation of any study-related procedures
* The subject and male partner must agree to participate in the infant follow-up if she becomes pregnant
* The subject must be able to communicate well with the investigator and research staff and to comply with the requirements of the study protocol.

Exclusion Criteria:

* ≥ four cumulus-oocyte-complexes (COCs) retrieved in a previous IVF cycles with a conventional stimulation protocol (within 6 months before enrollment)
* Serum value of FSH ≥25 IU/l (within 12 months measured in the absence of OC or hormone replacement intake)
* Thrombocytopenia defined as < 100.000 platelets/µl at screening
* Oral contraceptive or sex steroid intake within 1 month prior to enrollment
* Presence of structural or numerical chromosomal abnormality in cytogenetic analysis
* Relevant autoimmune disease
* History of malignancy and systemic chemotherapy or pelvic radiation
* Severe endometriosis (stage III-IV)
* Ovaries located outside the inner pelvis
* Presence of unilateral or bilateral hydrosalpinx
* Relevant endocrine disorders such as hypothalamic-pituitary disorder or thyroid dysfunction (except substituted Hashimoto's thyroiditis or latent hypothyroidism)
* Relevant thrombophilic disorder
* Contraindication for pregnancy
* Contraindication for transvaginal ovarian puncture (such as previous major lower abdominal surgery and known severe pelvic adhesion)
* Uterine malformations or pathologies (such as sub mucosal fibroid(s), endometrial hyperplasia, endometrial fluid accumulation, or endometrial adhesions)
* Mental disability or any other lack of fitness, in the investigator's opinion, to preclude subjects in or to complete the study

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 114 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Ovarian response | 34-36 hours following hCG administration at the end of ovarian stimulation
  Number of retrieved COCs per intention-to-treat

SECONDARY OUTCOMES:
Hormone levels | Follow-up period of three months entailing monthly evaluation
  Change from baseline in absolute and relative terms for Anti-Müllerian hormone (AMH), serum follicle stimulating hormone (FSH), luteinizing hormone (LH), estradiol (E2), testosterone (T) and antral follicle count (AFC)
Follicular response | On the day of triggering of final oocyte maturation or the day before
  Number of follicles (classified and summarised for every ovary as follows: mean diameter 10.0 - 11.9 mm, 12.0 - 13.9 mm, 14.0 - 15.9 mm, 16.0 - 17.9 mm, 18.0 - 19.9 mm and larger 19.9 mm)
COCs and MII oocytes | Day 0 after follicle puncture
  Mean number of retrieved COCs per protocol and mean number of metaphase II (MII) oocytes per protocol
Number of 2PN oocytes | Day 1 after follicle puncture
  Mean number per protocol
Mean number and quality of embryos | Day 2-5 after follicle puncture
  Grade a for cleavage stage embryo, >=3BB for blastocyst
Biochemical pregnancy rate | 12-16 days after oocyte pick-up
  Incidence of serum beta-hCG test > 25 mIU/ml per ITT and PP
Clinical pregnancy rate | 4 weeks after embryo transfer
  Incidence of gestational sac with heartbeat assessed by TVS per ITT and PP
Ongoing pregnancy rate | 8-10 weeks after embryo transfer
  Incidence of at least one foetus with heart beat assessed by TVS
Miscarriage rate | early (week 7-12 weeks of gestation); late (between 12 to 22 weeks of gestation)
  Defined as spontaneous loss of a clinical pregnancy rate, where embryo(s) or fetus(es) is/are nonviable and is/are not spontaneously absorbed or expelled from the uterus or surgically removed
Still birth rate | after 22 weeks of gestation
  Incidence of the delivery of a dead fetus
Live birth rate | at a follow-up time of 30 days after delivery
  Incidence of the birth of at least one live newborn after 22 weeks of gestation
Gestational age | at the day of delivery
  Gestational week estimated by calculating days from oocyte retrieval + 14 days
Weight of newborn | at the day of delivery
  Birth weight measured in gram
Length of newborn | at the day of delivery
  Birth length measured in centimeter
Incidence of birth sex | at the day of delivery
  Incidence of female or male newborn
Incidence of multiple birth | at the day of delivery
  Incidence of singleton/multiple newborns
Neonatal health | at a follow-up time of 30 days after delivery
  major and minor congenital anomalies
Post procedure pain | on the day of follicle puncture
  measured by a numerical rating scale from 0 (no pain) to 10 (worst pain)
Fertility Quality of Life Questionnaire | on the day of follicle puncture and embryo transfer
  FertiQoL International is a validated relational scale to assess the relational domain regarding quality of life in women undergoing infertility treatment. For each question, the patient will check the response that is closest to her current thoughts and feelings. Scale reaches depending on the question from "very dissatisfied" to "very satisfied", "always" to "never" or "an extreme amount" to "not at all".
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | at a follow-up time after 1, 2 and 5 years
  Incidence of adverse and serious adverse events with potential relationship to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Georg Griesing, MD, Principal Investigator — University of Luebeck
Locations (1):
- University of Luebeck, Lübeck, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will not be available before 2027
Access Criteria: reasonable request

REFERENCES:
- [Background] Gougeon A, Ecochard R, Thalabard JC. Age-related changes of the population of human ovarian follicles: increase in the disappearance rate of non-growing and early-growing follicles in aging women. Biol Reprod. 1994 Mar;50(3):653-63. doi: 10.1095/biolreprod50.3.653. PMID 8167237
- [Background] Martin JJ, Woods DC, Tilly JL. Implications and Current Limitations of Oogenesis from Female Germline or Oogonial Stem Cells in Adult Mammalian Ovaries. Cells. 2019 Jan 28;8(2):93. doi: 10.3390/cells8020093. PMID 30696098
- [Background] Maleki-Hajiagha A, Razavi M, Rouholamin S, Rezaeinejad M, Maroufizadeh S, Sepidarkish M. Intrauterine infusion of autologous platelet-rich plasma in women undergoing assisted reproduction: A systematic review and meta-analysis. J Reprod Immunol. 2020 Feb;137:103078. doi: 10.1016/j.jri.2019.103078. Epub 2019 Dec 31. PMID 32006776
- [Background] Sills ES, Rickers NS, Li X, Palermo GD. First data on in vitro fertilization and blastocyst formation after intraovarian injection of calcium gluconate-activated autologous platelet rich plasma. Gynecol Endocrinol. 2018 Sep;34(9):756-760. doi: 10.1080/09513590.2018.1445219. Epub 2018 Feb 28. PMID 29486615
- [Background] Danforth DR, Arbogast LK, Ghosh S, Dickerman A, Rofagha R, Friedman CI. Vascular endothelial growth factor stimulates preantral follicle growth in the rat ovary. Biol Reprod. 2003 May;68(5):1736-41. doi: 10.1095/biolreprod.101.000679. Epub 2002 Dec 11. PMID 12606430
- [Background] Quintana R, Kopcow L, Sueldo C, Marconi G, Rueda NG, Baranao RI. Direct injection of vascular endothelial growth factor into the ovary of mice promotes follicular development. Fertil Steril. 2004 Oct;82 Suppl 3:1101-5. doi: 10.1016/j.fertnstert.2004.03.036. PMID 15474081
- [Background] Bakacak M, Bostanci MS, Inanc F, Yaylali A, Serin S, Attar R, Yildirim G, Yildirim OK. Protective Effect of Platelet Rich Plasma on Experimental Ischemia/Reperfusion Injury in Rat Ovary. Gynecol Obstet Invest. 2016;81(3):225-31. doi: 10.1159/000440617. Epub 2015 Oct 24. PMID 26496072
- [Background] Ozcan P, Takmaz T, Tok OE, Islek S, Yigit EN, Ficicioglu C. The protective effect of platelet-rich plasma administrated on ovarian function in female rats with Cy-induced ovarian damage. J Assist Reprod Genet. 2020 Apr;37(4):865-873. doi: 10.1007/s10815-020-01689-7. Epub 2020 Feb 4. PMID 32020412
- [Background] Atkinson L, Martin F, Sturmey RG. Intraovarian injection of platelet-rich plasma in assisted reproduction: too much too soon? Hum Reprod. 2021 Jun 18;36(7):1737-1750. doi: 10.1093/humrep/deab106. PMID 33963408
- [Background] Melo P, Navarro C, Jones C, Coward K, Coleman L. The use of autologous platelet-rich plasma (PRP) versus no intervention in women with low ovarian reserve undergoing fertility treatment: a non-randomized interventional study. J Assist Reprod Genet. 2020 Apr;37(4):855-863. doi: 10.1007/s10815-020-01710-z. Epub 2020 Feb 7. PMID 32030554
- [Background] Urman B, Boza A, Balaban B. Platelet-rich plasma another add-on treatment getting out of hand? How can clinicians preserve the best interest of their patients? Hum Reprod. 2019 Nov 1;34(11):2099-2103. doi: 10.1093/humrep/dez190. PMID 31725883
- [Background] Farimani M, Heshmati S, Poorolajal J, Bahmanzadeh M. A report on three live births in women with poor ovarian response following intra-ovarian injection of platelet-rich plasma (PRP). Mol Biol Rep. 2019 Apr;46(2):1611-1616. doi: 10.1007/s11033-019-04609-w. Epub 2019 Feb 5. PMID 30725347
- [Background] Sills ES, Wood SH. Autologous activated platelet-rich plasma injection into adult human ovary tissue: molecular mechanism, analysis, and discussion of reproductive response. Biosci Rep. 2019 Jun 4;39(6):BSR20190805. doi: 10.1042/BSR20190805. Print 2019 Jun 28. PMID 31092698
- [Background] Hsu CC, Hsu L, Hsu I, Chiu YJ, Dorjee S. Live Birth in Woman With Premature Ovarian Insufficiency Receiving Ovarian Administration of Platelet-Rich Plasma (PRP) in Combination With Gonadotropin: A Case Report. Front Endocrinol (Lausanne). 2020 Feb 19;11:50. doi: 10.3389/fendo.2020.00050. eCollection 2020. PMID 32140135